CLINICAL TRIAL: NCT01846650
Title: A Bioequivalence Study of Capecitabine Tablets in Patients of Locally Advanced or Metastatic Breast Cancer or Metastatic Colorectal Cancer
Brief Title: A Bioequivalence Study of Capecitabine Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KPTB-1.1
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Metastatic Breast Cancer or Metastatic Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine tablets (Experimental): Single oral Capecitabine tablets 2000mg qd
  Interventions: Drug: Capecitabine tablets
- XELODA (Active Comparator): Single oral XELODA 2000mg qd
  Interventions: Drug: XELODA

INTERVENTIONS:
Drug: Capecitabine tablets — Single oral Capecitabine tablets 2000mg qd
  Arms: Capecitabine tablets
Drug: XELODA — Single oral XELODA 2000mg qd
  Arms: XELODA

SUMMARY:
1. purpose: To conduct the relative bioavalability study of Capecitabine tablets 500 mg (Jiangsu Chia-Tai Tianqing Pharmacy Co. Ltd.) versus XELODA® 500 mg tablets (Manufactured by Roche Pharma AG)
2. Experimental Design： Two-period crossover design
3. Test drug: Capecitabine tablets Reference drug: XELODA
4. Sample size：24

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathologically /cytologically confirmed breast cancer or colorectal cancer，without chemotherapy or only adjuvant chemotherapy, and had previously received one or two standard chemotherapy regimens for patients;
* Age: 18-70 years, gender: both，BMI≥17，Eastern Cooperative Oncology Group (ECOG) performance status：0-2，Life expectancy greater than 3 months;
* Patients must have normal bone marrow function, liver and kidney function; adequate organ function in the last 1 week, meeting the following: ANC≥1.5×109/L，PLT≥80×109/L, Total bilirubin≤1.5×the upper limit of normal, ALT,AST≤2.5×the upper limit of normal, creatinine≤1.5×the institutional upper limit of normal.
* Patients who has retreatment could be enrolled at least 4 weeks after the last chemotherapy and radiotherapy.
* Patients must volunteer to participate and sign informed consent form.

Exclusion Criteria:

* Suffering from heart, liver, kidney disease or severe acute and Organ invasion disease;
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil, or known DPD (Dihydropyrimidine Dehydrogenase) deficiency.
* Pregnant or breast-feeding female
* Only bone metastasis lesions, no other measurable lesions
* Known brain metastasis or history of organ transplantation
* Have long-term systemic steroid therapy
* Serious diseases of vital organs; other malignancies which is not cure
* Use of chemotherapy in the last 4 weeks
* History of drug/alcohol addiction or a positive hepatitis screen including hepatitis B surface antigen, HCV or HAV (IgM) antibodies
* Patient having abnormal serum calcium level at screening visit which as judged by Investigator could lead to safety risk to the patient upon participation in the trial or could interfere with the conduct of the trial.
* Pre-existing motor or sensory neurotoxicity of a severity grade 2 by NCI CTCAE criteria or known, existing uncontrolled coagulopathy.
* Subjects are thought unsuitable for the study by investigators;
* Inability to comply with protocol or study procedures in the opinion of the investigator;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | predose, 0.33,0.67，1,1.5,2，2.5，3,4，5,6，8,hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ai dong, doctor, Principal Investigator — First Affiliated Hospital of Fourth Military Medical University
Locations (1):
- First Affiliated Hospital of Fourth Military Medical University, Xi’an, Shanxi, China